CLINICAL TRIAL: NCT04265586
Title: Sleep, Pain and Health-related Quality of Life in Chronic Pain Patients. Interventional Study
Brief Title: Sleep, Pain and Quality of Life in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Reetta Sipilä, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/577/2019
Record Dates: First submitted 2020-01-24; First posted 2020-02-11 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain; Insomnia
Keywords: Health-related Quality of Life; Anxiety; Pain intensity; Pain interference; Symptoms of insomnia
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Pain | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No insomnia (No Intervention): This group contains participants who report only mild symptoms of insomnia (Insomnia Severity Index, ISI<15).
- Digital Cognitive Behavioural Therapy (iCBT) (Experimental): This group contains participants with moderate to severe symptoms of insomnia symptoms (Insomnia Severity Index, ISI >14). Intervention is iCBT for participants with insomnia (7-16 weeks).
  Interventions: Behavioral: Web-based Cognitive Behavioural Therapy (iCBT)
- Sleep hygiene education (Experimental): This group contains participants with moderate to severe symptoms of insomnia symptoms (Insomnia Severity Index, ISI >14). Sleep hygiene education (approximately 1 hour)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Sleep hygiene education is either face-to-face appointment or "video-meeting" with trained nurse.
  Arms: Sleep hygiene education
Behavioral: Web-based Cognitive Behavioural Therapy (iCBT) — iCBT is a web-based programme (7-16 weeks) designed to treat the symptoms of insomnia.
  Arms: Digital Cognitive Behavioural Therapy (iCBT)

SUMMARY:
The interventional study will have two main aims. First, to compare two interventions aiming to improve sleep in chronic pain patients. And secondly, to study the associations of sleep, mood, chronic pain and quality of life. Half of participants will go through iCBT intervention for insomnia and the other half will receive sleep hygiene education. Additionally, the study will gather information which patients will benefit/will not benefit the tertiary pain clinic treatment when the outcome variable is the Health-related Quality of Life (HrQoL).

DETAILED DESCRIPTION:
Sleep disturbances associates closely with chronic pain. It now seems that sleep problems usually precede and maintain persistent pain. Anxiety and worry frequently precede and associate with disturbed sleep and chronic pain. Depression is usually a consequence of chronic pain. Pain and depression disturb sleep further. These elements form a vicious circle where poor sleep is a critical driver.

Previous studies have shown that sleep disturbances are a major contributor to the poor health-related quality of life (HRQoL) of patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* fluency in Finnish

Exclusion Criteria:

* severe psychiatric conditions (e.g. scizopherenia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life (HrQoL) questionnaire (15D) | Change from Baseline HrQoL at 12 months
  15-item questionnaire of HrQoL, ranging from 15 to 75 smaller value indicates better HrQoL

SECONDARY OUTCOMES:
Mood -BDI-II and STAI-Y | Change from Baseline mood at 12 months
  Questionnaires about depression and anxiety, BDI-II values ranging from 0-63, and STAI-Y values ranging form 20-80 for both state and trait anxiety. Higher values in both questionnaires indicates higher amount of asked symptom.
Pain related catastrophizing (PCS) | Change from Baseline pain related catatsrophizing at 12 months
  Pain catastrophizing Scale, values ranging from 0 to 52, higher values indicating higher catasrophizing tendency.
Stress and worrying tendency | Change from Baseline stress and worrying tendency at 12 months
  Questionnaires about perceived stress and worrying tendency. Values ranges from 16 to 80, higher values indicating higher amount of worring tendency.
Brief Pain Inventory (BPI) | Change from Baseline pain intensity and interference at 12 months
  12-item questionnaire abour self-reported pain intensity and interference. Values ranges from 0 to 120, higher values indicating higher amount of pain interference and intensity.
Insomnia Severity Index (ISI) | Change from Baseline symptoms of insomnia at 12 months
  5-item questionnaire of self-reported symptoms of insomnia. Values ranging from 0 to 28, higher values indicating higer amount of symptoms of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Eija A Kalso, Professor, Principal Investigator — Helsinki University Hospital, University of Helsinki
Locations (2):
- Finland (2):
  - HUH Pain Clinic, Helsinki
  - Turku University Hospitla Pain Clinic, Turku

IPD SHARING:
Plan to Share IPD: No